CLINICAL TRIAL: NCT05099640
Title: A Phase 3 Study of PTC923 in Subjects With Phenylketonuria
Brief Title: A Study of PTC923 in Participants With Phenylketonuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC923-MD-003-PKU; 2021-000474-29 (EudraCT Number)
Record Dates: First submitted 2021-10-06; First posted 2021-10-29 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: PTC923 (Experimental): Participants will receive PTC923 7.5 milligrams (mg)/kilogram (kg) (participants 0 to <6 months of age), 15 mg/kg (participants 6 to <12 months of age), 30 mg/kg (participants 12 months to <2 years of age), or 60 mg/kg (participants ≥2 years of age) orally once daily for 14 days.
  Interventions: Drug: PTC923
- Part 2: PTC923 (Experimental): Participants will receive PTC923 20 mg/kg daily for Weeks 1 and 2, then PTC923 40 mg/kg daily for Weeks 3 and 4, then PTC923 60 mg/kg daily for Weeks 5 and 6.
  Interventions: Drug: PTC923
- Part 2: Placebo (Placebo Comparator): Participants will receive equivalent quantities of placebo to match the 20 to 40 to 60 mg/kg dose escalation of the PTC923 treatment arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTC923 — PTC923 powder for oral use will be suspended in water or apple juice prior to administration.
  Arms: Part 1: PTC923; Part 2: PTC923
Drug: Placebo — Placebo matching to PTC923
  Arms: Part 2: Placebo

SUMMARY:
The main purpose of this trial is to evaluate the efficacy of PTC923 in reducing blood phenylalanine (Phe) levels in participants with phenylketonuria as measured by mean change in blood Phe levels from baseline to Weeks 5 and 6 (that is, the average of each respective treatment dose 2-week period of double-blind treatment).

DETAILED DESCRIPTION:
The study includes 2 parts: Part 1 and 2. Part 1 of the study tests for responsiveness to PTC923, with 14 days of open-label treatment with PTC923. At the end of treatment in Part 1, the mean change in blood Phe levels over the 14-day treatment period for all participants will be assessed against their pretreatment (baseline) blood Phe level. Participants ≥2 years of age who experience a <15% reduction in blood Phe levels will be classified as non-responsive and participation in the study will be terminated. Participants (≥2 years of age) who experience a ≥15% reduction in blood Phe levels will continue into Part 2. Participants <2 years of age who experience ≥15% reduction in blood Phe levels will be offered the option to enroll directly into an open-label extension Study PTC923-MD-004-PKU. Participants <2 years of age who experience a <15% reduction in blood Phe levels will be classified as nonresponsive, and participation in the study will be terminated. Following the minimum 14-day PTC923 washout period, all eligible participants will be randomized in Part 2 to receive either PTC923 or placebo. After 6 weeks of treatment with either PTC923 or placebo, participants will be offered the option to enter an open-label extension Study PTC923-MD-004-PKU (NCT05166161).

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled blood Phe level ≥360 μmol/L on current therapy anytime during screening and uncontrolled blood Phe level ≥360 μmol/L on current therapy when taking the average of the 3 most recent Phe levels from the participant's medical history (inclusive of the screening value).
* Clinical diagnosis of phenylketonuria with hyperphenylalaninemia (HPA) documented by past medical history of at least 2 blood Phe measurements ≥600 μmol/L.
* Women of childbearing potential must have a negative pregnancy test at screening and agree to abstinence or the use of at least one highly effective form of contraception for the duration of the study, and for up to 90 days after the last dose of study drug.
* Males who are sexually active with women of childbearing potential who have not had a vasectomy must agree to use a barrier method of birth control during the study and for up to 90 days after the last dose of study drug. Males must also refrain from sperm donations during this time period.
* Willing to continue current diet unchanged while participating in the study.

Exclusion Criteria:

* Gastrointestinal disease (such as irritable bowel syndrome, inflammatory bowel disease, chronic gastritis, and peptic ulcer disease, etc.) that could affect the absorption of study drug.
* History of gastric surgery, including Roux-en-Y gastric bypass surgery or an antrectomy with vagotomy, or gastrectomy.
* History of allergies or adverse reactions to synthetic tetrahydrobiopterin (BH4) or sepiapterin.
* Current participation in any other investigational drug study or use of any investigational agent within 30 days prior to screening.
* Any clinically significant laboratory abnormality as determined by the investigator.
* A female who is pregnant or breastfeeding, or considering pregnancy.
* Serious neuropsychiatric illness (for example, major depression) not currently under medical control, that in the opinion of the investigator or sponsor, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant.
* Past medical history and/or evidence of renal impairment and/or condition including moderate/severe renal insufficiency (glomerular filtration rate [GFR] <60 milliliters [mL]/minute [min]) and/or under care of a nephrologist.
* Any abnormal physical examination and/or laboratory findings indicative of signs or symptoms of renal disease, including calculated GFR <60 mL/min/1.73 square meter (m^2).
* Requirement for concomitant treatment with any drug known to inhibit folate synthesis (for example, methotrexate).
* Confirmed diagnosis of a primary BH4 deficiency as evidenced by biallelic pathogenic mutations in 6-pyruvoyltetrahydropterin synthase, recessive guanosine-5'-triphosphate (GTP) cyclohydrolase I, sepiapterin reductase, quinoid dihydropteridine reductase, or pterin-4-alpha-carbinolamine dehydratase genes.
* Major surgery within the prior 90 days of screening.
* Concomitant treatment with BH4 supplementation (for example, sapropterin dihydrochloride, KUVAN) or pegvaliase-pqpz (PALYNZIQ).
* Unwillingness to washout from BH4 supplementation (for example, sapropterin dihydrochloride, KUVAN) or pegvaliase-pqpz (PALYNZIQ)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (12):
  - Stanford University Center for Academic Medicine, Stanford, California
  - University of Colorado and the Children's Hospital CO, Aurora, Colorado
  - UF College of Medicine, Department of Pediatrics Division of Genetics and Metabolism, Gainesville, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai (ISMMS), New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Texas Health Science Center of Texas, Houston, Texas
  - University of Utah, Division of Medical Genetics (pediatric and adult clinic), Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Westmead Hospital, Westmead, New South Wales
  - PARC Clinical Research, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
- Brazil (2):
  - Hospital de clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo
- Canada (2):
  - Metabolics and Genetics in Calgary (MAGIC) Clinic, Ltd., Calgary, Alberta
  - The Hospital for Sick Children University of Toronto, Adult Clinic: The Fred A Litwin Family Centre in Genetic Medicine University Health Network & Mt. Sinai Hospital, Toronto, Ontario
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Bretonneau Hospital - CHRU de Tours, Tours, Centre-Val de Loire
  - CHRU de Tours- Hôpital Pédiatrique de Clocheville, Tours, Centre-Val de Loire
- Pediatric Surgery Center, Tbilisi, Georgia
- Germany (3):
  - University Children's Hospital Hamburg Eppendorf (Kinder-UKE) Klinik für Kinder- und Jugendmedizin (Kinder-UKE), Hamburg
  - Universitätsklinikum Heidelberg / Zentrum für Kinder- und Jugendmedizin / Sektion für Neuropädiatrie & Stoffwechselmedizin, Heidelberg
  - Universitätsklinikum Münster, Münster
- Italy (2):
  - Policlinico Umberto I, Rome, Lazio
  - Division of Inherited Metabolic Diseases, Azienda Ospedaliera-Università Padova, Padua, Veneto
- Mexico (2):
  - PanAmerican Clinical Research, Guadalajara, Jalisco
  - Grupo Médico Camino SC, Benito Juárez, Mexico City
- UMCG Beatrix Children's Hospital, Groningen, Netherlands
- Portugal (3):
  - Centro Hospitalar Universitário Do Porto, Epe, Porto, Douro Litoral
  - CENTRO HOSPITALAR UNIVERSITÁRIO LISBOA NORTE Hospital de Santa Maria,, Lisbon, Estremadura
  - CENTRO HOSPITALAR UNIVERSITÁRIO LISBOA NORTE Hospital de Santa Maria, Lisbon, Estremadura
- Spain (2):
  - Hospital Sant Joan de Déu, Barcelona, Esplugues de Llobregat
  - Hospital Universitario Ramón y Cajal, Madrid
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Altındağ, Ankara
  - Gazi Üniversitesi Tıp Fakültesi, Yenimahalle, Ankara
  - İstanbul Üniversitesi Cerrahpaşa Tıp Fakültesi, Fatih, Istanbul
  - Ege University Faculty of Medicine Children Hospital, Bornova, İzmir
  - Cukurova Üniversity Balcali Hospital Health Application and Research Center, Adana
- United Kingdom (2):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Great Ormond Street Hospital, London

REFERENCES:
- [Derived] Muntau AC, Gallagher S, Lah M, Belanger-Quintana A, Longo N. Sepiapterin as a treatment for people living with phenylketonuria: a plain language summary of the APHENITY trial. J Comp Eff Res. 2026 Jan;15(1):e250116. doi: 10.57264/cer-2025-0116. Epub 2025 Dec 9. PMID 41363942
- [Derived] Muntau AC, Longo N, Ezgu F, Schwartz IVD, Lah M, Bratkovic D, Margvelashvili L, Kiykim E, Zori R, Campistol Plana J, Belanger-Quintana A, Lund A, Guilder L, Chakrapani A, Mungan HN, Guimas A, Cabrales Guerra IDC, MacDonald A, Ingalls K, Smith N; APHENITY study group. Effects of oral sepiapterin on blood Phe concentration in a broad range of patients with phenylketonuria (APHENITY): results of an international, phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2024 Oct 5;404(10460):1333-1345. doi: 10.1016/S0140-6736(24)01556-3. PMID 39368841

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts: Part 1: Open-label and Part 2: Placebo-controlled Randomized Treatment. In Part 1, 157 participants received sepiapterin. In Part 2, 56 participants received sepiapterin and 54 participants received placebo.
Pre-assignment Details: Participants (≥2 years of age) who experienced a ≥15% reduction in blood Phe levels (responder) continued into Part 2. Non-responders did not continue to Part 2.
Groups:
- Part 1: Sepiapterin: Participants received sepiapterin 30 milligrams (mg)/kilogram (kg) (participants 12 months to <2 years of age) or 60 mg/kg (participants ≥2 years of age) orally once daily for 14 days.
- Part 2: Sepiapterin: Participants received sepiapterin 20 mg/kg daily for Weeks 1 and 2, then sepiapterin 40 mg/kg daily for Weeks 3 and 4, then sepiapterin 60 mg/kg daily for Weeks 5 and 6.
- Part 2: Placebo: Participants received equivalent quantities of placebo to match the 20 to 40 to 60 mg/kg dose escalation of the sepiapterin treatment arm.
Period: Part 1: Open-label (14 Days)
Arm/Group | Part 1: Sepiapterin | Part 2: Sepiapterin | Part 2: Placebo
Started | 157 | 0 | 0
Received at Least 1 Dose of Study Drug | 157 | 0 | 0
Completed | 111 (110 participants were eligible to progress to Part 2.) | 0 | 0
Not Completed | 46 | 0 | 0
Not completed — Non-responsive for sepiapterin | 39 | 0 | 0
Not completed — Participant decision | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Other than specified | 2 | 0 | 0
Period: Part 2: Randomized Treatment (6 Weeks)
Arm/Group | Part 1: Sepiapterin | Part 2: Sepiapterin | Part 2: Placebo
Started | 0 | 56 | 54
Received at Least 1 Dose of Study Drug | 0 | 56 | 54
Completed | 0 | 55 | 54
Not Completed | 0 | 1 | 0
Not completed — Participant decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug, including during Part 1. Part 2 included participants (≥2 years of age) who experienced a ≥15% reduction in blood Phe levels (responder). Non-responders in Part 1 did not continue to Part 2.
Groups:
- Part 1 (Participants Who Participated in Part 1 Only): Sepiapterin: Participants received sepiapterin 30 mg/kg (participants 12 months to <2 years of age) or 60 mg/kg (participants ≥2 years of age) orally once daily for 14 days.
- Total: Total of all reporting groups
Arm/Group | Part 1 (Participants Who Participated in Part 1 Only): Sepiapterin | Part 2: Sepiapterin | Part 2: Placebo | Total
Number analyzed (Participants) | 47 | 56 | 54 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.4 (15.07) | 16.5 (11.12) | 18.4 (10.65) | 17.7 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 27 | 72
  Male | 28 | 30 | 27 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 12 | 25
  Not Hispanic or Latino | 40 | 47 | 42 | 129
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 2 | 8
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 41 | 52 | 49 | 142
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 3 | 7
Blood Phenylketonuria (Phe) Level [Mean (Standard Deviation); unit: micromoles (μmol)/liter (L)] — Population: Baseline blood Phe level data is reported for Part 1 and Part 2 separately in different rows.
  micromoles (μmol)/liter (L)
    Part 1 (Participants who Participated in Part 1 Only) (Non-responders): number analyzed (Participants) | 47 | 0 | 0 | 47
    Part 1 (Participants who Participated in Part 1 Only) (Non-responders) | 651.16 (333.439) |  |  | 651.16 (333.439)
    Part 2 (Randomized Responders from Part 1): number analyzed (Participants) | 0 | 56 | 54 | 110
    Part 2 (Randomized Responders from Part 1) |  | 645.59 (246.085) | 667.81 (264.574) | 656.50 (254.397)
Blood Phe Level in Classical PKU Participants [Mean (Standard Deviation); unit: μmol/L] — Classical PKU participants: Participants with severe forms of PKU, typically had very high blood Phe levels (>1200 μmol/L). Population: Baseline blood Phe level data is reported for Part 1 and Part 2 classical PKU participants separately in different rows.
  μmol/L
    Part 1 (Participants who Participated in Part 1 Only) (Non-responders with Classical PKU): number analyzed (Participants) | 17 | 0 | 0 | 17
    Part 1 (Participants who Participated in Part 1 Only) (Non-responders with Classical PKU) | 1495.8 (641.18) |  |  | 1495.8 (641.18)
    Part 2 (Randomized Responders from Part 1 with Classical PKU): number analyzed (Participants) | 0 | 8 | 11 | 19
    Part 2 (Randomized Responders from Part 1 with Classical PKU) |  | 737.56 (277.279) | 812.14 (295.239) | 780.74 (282.411)

OUTCOME MEASURES:

1. Primary Outcome: Part 2 Double-blind Phase: Mean Change From Baseline in Blood Phenylketonuria (Phe) Level to Weeks 5 and 6 (Averaged Over a 2-week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 2, and mean level at Weeks 5 and 6 was calculated as the average of blood Phe levels collected during the Week 5-6 analysis visit window. Least square (LS) mean and standard error (SE) were calculated using mixed model repeated measures (MMRM) method.
Time Frame: Baseline, Weeks 5 and 6 (average of the 2-week period)
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = participants of FAS with Phe reduction from Baseline ≥30% during Part 1, who continued in Part 2. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 49 | 49
μmol/L | -415.75 (24.066) | -19.88 (24.223)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -395.87, 95% CI 2-sided [-463.07 to -328.66], Standard Error of Mean 33.848

2. Primary Outcome: Part 2 Double-blind Phase: Percent Change From Baseline in Blood Phe Level to Weeks 5 and 6 (Averaged Over a 2-week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 2, and mean level at Weeks 5 and 6 was calculated as the average of blood Phe levels collected during the Week 5-6 analysis visit window. LS mean and SE were calculated using MMRM method.
Time Frame: Baseline, Weeks 5 and 6 (average of the 2-week period)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = participants of FAS with Phe reduction from Baseline ≥30% during Part 1, who continued in Part 2. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 49 | 49
percent change | -63.40 (3.537) | 0.82 (3.561)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -64.22, 95% CI 2-sided [-74.09 to -54.35], Standard Error of Mean 4.973

3. Secondary Outcome: Part 2 Double-blind Phase: Percentage of Participants With Baseline Phe Levels ≥600 μmol/L Who Achieved Phe Levels <600 μmol/L in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 2, and mean level at Weeks 5 and 6 was calculated as the average of blood Phe levels collected during the Week 5-6 analysis visit window.
Time Frame: Weeks 5 and 6 (average of the 2-week period)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = participants of FAS with Phe reduction from baseline ≥30% during Part 1 and had Part 2 baseline Phe levels ≥600 μmol/L. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 28 | 30
percentage of participants | 92.9 [76.50 to 99.12] | 30.0 [14.73 to 49.40]
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Chi-squared; Odds Ratio (OR) = 30.33, 95% CI 2-sided [5.30 to 294.24]

4. Secondary Outcome: Part 2 Double-blind Phase: Percentage of Participants With Baseline Phe Levels ≥360 μmol/L Who Achieved Phe Levels <360 μmol/L in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: as for outcome 3
Time Frame: Weeks 5 and 6 (average of the 2-week period)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = participants of FAS with Phe reduction from baseline ≥30% during Part 1 and Part 2 baseline Phe levels ≥360 μmol/L. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 44 | 43
percentage of participants | 84.1 [69.93 to 93.36] | 9.3 [2.59 to 22.14]
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Chi-squared; Odds Ratio (OR) = 51.54, 95% CI 2-sided [12.28 to 245.34]

5. Secondary Outcome: Part 2 Double-blind Phase: Mean Change From Baseline in Blood Phe Level at Each 2-Week Period (Averaged Over Each 2-Week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 2, and mean levels at Weeks 1 and 2, Weeks 3 and 4, and Weeks 5 and 6 were calculated as the average of blood Phe levels collected during the Week 1-2, Week 3-4, and Week 5-6 analysis visit windows, respectively.
Time Frame: Baseline, Weeks 1 and 2, Weeks 3 and 4, and Weeks 5 and 6 (average of each 2-week period)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = participants of FAS with Phe reduction from Baseline ≥30% during Part 1 and continued in Part 2. 'Number analyzed' = participants evaluable at specified timepoint. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 49 | 49
μmol/L
  Weeks 1 and 2 | -341.18 (226.178) | -53.27 (174.461)
  Weeks 3 and 4: number analyzed (Participants) | 49 | 48
  Weeks 3 and 4 | -406.88 (199.259) | -30.43 (203.425)
  Weeks 5 and 6 | -410.07 (204.442) | -16.19 (198.642)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 1 and 2: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -289.89, 95% CI 2-sided [-356.29 to -223.50], Standard Error of Mean 33.440
Statistical Analysis 2: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 3 and 4: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -375.47, 95% CI 2-sided [-435.88 to -315.06], Standard Error of Mean 30.424
Statistical Analysis 3: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 5 and 6: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -395.87, 95% CI 2-sided [-463.07 to -328.66], Standard Error of Mean 33.848

6. Secondary Outcome: Part 2 Double-blind Phase: Percent Change From Baseline in Blood Phe Level at Each 2-Week Period (Averaged Over Each 2-Week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: as for outcome 5
Time Frame: Baseline, Weeks 1 and 2, Weeks 3 and 4, and Weeks 5 and 6 (average of each 2-week period)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 49 | 49
percent change
  Weeks 1 and 2 | -48.55 (4.265) | -6.04 (4.285)
  Weeks 3 and 4: number analyzed (Participants) | 49 | 48
  Weeks 3 and 4 | -62.46 (3.220) | -1.43 (3.257)
  Weeks 5 and 6 | -63.40 (3.537) | 0.82 (3.561)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 1 and 2: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -42.52, 95% CI 2-sided [-54.45 to -30.59], Standard Error of Mean 6.008
Statistical Analysis 2: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 3 and 4: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -61.03, 95% CI 2-sided [-70.02 to -52.03], Standard Error of Mean 4.531
Statistical Analysis 3: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Weeks 5 and 6: Sepiapterin vs. Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -64.22, 95% CI 2-sided [-74.09 to -54.35], Standard Error of Mean 4.973

7. Secondary Outcome: Part 1 Open-label Run-in Phase: Plasma Concentration of Tetrahydrobiopterin (BH4) and Sepiapterin
Time Frame: Predose, 0.5, 1, 2, 4, 6, 8, and 24 hours postdose at Day 1; 2 and 6 hours postdose at Day 14
Population: Pharmacokinetic (PK) Analysis Set included all participants who had at least 1 measurable plasma concentration of sepiapterin or BH4. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/milliliter (mL)
Groups:
- Part 1: Sepiapterin: Participants received sepiapterin 30 mg/kg (participants 12 months to <2 years of age) or 60 mg/kg (participants ≥2 years of age) orally once daily for 14 days.
Arm/Group | Part 1: Sepiapterin
Number analyzed (Participants) | 17
nanograms (ng)/milliliter (mL)
  BH4: Day 1 (predose): number analyzed (Participants) | 16
  BH4: Day 1 (predose) | 10.6 (5.34)
  BH4: Day 1 (0.5 hr): number analyzed (Participants) | 16
  BH4: Day 1 (0.5 hr) | 22.3 (13.2)
  BH4: Day 1 (1 hr): number analyzed (Participants) | 15
  BH4: Day 1 (1 hr) | 107 (76.0)
  BH4: Day 1 (2 hrs): number analyzed (Participants) | 16
  BH4: Day 1 (2 hrs) | 236 (124)
  BH4: Day 1 (4 hrs): number analyzed (Participants) | 16
  BH4: Day 1 (4 hrs) | 289 (170)
  BH4: Day 1 (6 hrs): number analyzed (Participants) | 14
  BH4: Day 1 (6 hrs) | 245 (131)
  BH4: Day 1 (8 hrs): number analyzed (Participants) | 15
  BH4: Day 1 (8 hrs) | 205 (130)
  BH4: Day 1 (24 hrs): number analyzed (Participants) | 16
  BH4: Day 1 (24 hrs) | 25.5 (21.1)
  BH4: Day 14 (2 hrs): number analyzed (Participants) | 1
  BH4: Day 14 (2 hrs) | 94.1
  BH4: Day 14 (6 hrs): number analyzed (Participants) | 1
  BH4: Day 14 (6 hrs) | 105
  Sepiapterin: Day 1 (predose): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (predose) | 0.000 (0.000)
  Sepiapterin: Day 1 (0.5 hr): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (0.5 hr) | 0.939 (0.940)
  Sepiapterin: Day 1 (1 hr): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (1 hr) | 2.22 (1.11)
  Sepiapterin: Day 1 (2 hrs): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (2 hrs) | 2.06 (1.10)
  Sepiapterin: Day 1 (4 hrs) | 1.73 (1.58)
  Sepiapterin: Day 1 (6 hrs): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (6 hrs) | 1.60 (2.13)
  Sepiapterin: Day 1 (8 hrs): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (8 hrs) | 0.493 (0.598)
  Sepiapterin: Day 1 (24 hrs): number analyzed (Participants) | 16
  Sepiapterin: Day 1 (24 hrs) | 0.436 (0.987)
  Sepiapterin: Day 14 (2 hrs): number analyzed (Participants) | 1
  Sepiapterin: Day 14 (2 hrs) | 3.33
  Sepiapterin: Day 14 (6 hrs): number analyzed (Participants) | 1
  Sepiapterin: Day 14 (6 hrs) | 2.82

8. Secondary Outcome: Part 2 Double-blind Phase: Plasma Concentration of BH4 and Sepiapterin
Time Frame: Predose and 4 hours postdose at Days 1, 14, 28, and 42
Population: PK Analysis Set included all participants who had at least 1 measurable plasma concentration of sepiapterin or BH4. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 4 | 4
ng/mL
  BH4: Day 1 (predose): number analyzed (Participants) | 4 | 2
  BH4: Day 1 (predose) | 6.63 (3.60) | 8.52 (4.36)
  BH4: Day 1 (4 hrs): number analyzed (Participants) | 3 | 4
  BH4: Day 1 (4 hrs) | 351 (184) | 12.4 (1.74)
  BH4: Day 14 (predose): number analyzed (Participants) | 4 | 3
  BH4: Day 14 (predose) | 7.04 (3.13) | 4.27 (4.93)
  BH4: Day 14 (4 hrs): number analyzed (Participants) | 2 | 4
  BH4: Day 14 (4 hrs) | 401 (184) | 11.3 (8.70)
  BH4: Day 28 (predose): number analyzed (Participants) | 3 | 4
  BH4: Day 28 (predose) | 11.8 (6.29) | 9.70 (4.18)
  BH4: Day 28 (4 hrs): number analyzed (Participants) | 3 | 4
  BH4: Day 28 (4 hrs) | 406 (57.5) | 12.2 (4.46)
  BH4: Day 42 (predose) | 10.0 (6.43) | 9.41 (4.58)
  BH4: Day 42 (4 hrs): number analyzed (Participants) | 2 | 4
  BH4: Day 42 (4 hrs) | 442 (197) | 11.4 (3.91)
  Sepiapterin: Day 1 (predose) | 0.000 (0.000) | 0.000 (0.000)
  Sepiapterin: Day 1 (4 hrs): number analyzed (Participants) | 3 | 4
  Sepiapterin: Day 1 (4 hrs) | 0.620 (1.07) | 0.000 (0.000)
  Sepiapterin: Day 14 (predose): number analyzed (Participants) | 4 | 3
  Sepiapterin: Day 14 (predose) | 0.000 (0.000) | 0.000 (0.000)
  Sepiapterin: Day 14 (4 hrs): number analyzed (Participants) | 3 | 4
  Sepiapterin: Day 14 (4 hrs) | 1.23 (1.26) | 0.000 (0.000)
  Sepiapterin: Day 28 (predose): number analyzed (Participants) | 4 | 3
  Sepiapterin: Day 28 (predose) | 0.000 (0.000) | 0.000 (0.000)
  Sepiapterin: Day 28 (4 hrs): number analyzed (Participants) | 3 | 4
  Sepiapterin: Day 28 (4 hrs) | 1.17 (1.09) | 0.000 (0.000)
  Sepiapterin: Day 42 (predose) | 0.000 (0.000) | 0.000 (0.000)
  Sepiapterin: Day 42 (4 hrs): number analyzed (Participants) | 3 | 4
  Sepiapterin: Day 42 (4 hrs) | 1.03 (1.14) | 0.000 (0.000)

9. Secondary Outcome: Part 1 Open-label Run-in Phase: Area Under the Concentration-time Curve From Time 0 to 24 Hours Postdose (AUC0-24h) of Sepiapterin and BH4 Following the First Dose of Sepiapterin at 60 mg/kg
Time Frame: 0 to 24 hours postdose at Day 1
Population: PK Analysis Set included all participants who had at least 1 measurable plasma concentration of sepiapterin or BH4. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Part 1: Sepiapterin
Number analyzed (Participants) | 16
hours*ng/mL
  BH4 | 2990 (1450)
  Sepiapterin | 19.6 (20.1)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs were considered:
  * Part 1 TEAEs, which included all AEs occurring after first dose in Part 1 but before first dose in Part 2;
  * Part 2 TEAEs, which included all AEs after first randomized dose in Part 2. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Day 42
Population: Safety analysis set included all participants who received at least 1 dose of study drug, including during Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Sepiapterin | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 157 | 56 | 54
Participants | 68 | 33 | 18

11. Other Pre Specified Outcome: Part 2 Double-blind Phase: Mean Change From Baseline in Blood Phe Level to Weeks 5 and 6 (Averaged Over a 2-week Period) in Classical PKU Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Classical PKU participants: Participants with severe forms of PKU, typically very high blood Phe levels (>1200 μmol/L). Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 2, and mean level at Weeks 5 and 6 was calculated as the average of blood Phe levels collected during the Week 5-6 analysis visit window. LS mean and SE were calculated using MMRM method.
Time Frame: Baseline, Weeks 5 and 6 (average of the 2-week period)
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study drug in Part 2. Non-responders in Part 1 did not continue to Part 2 and were not included in the analysis. Here, 'Overall number of participants analyzed' = Classical PKU participants of FAS with Phe reduction from Baseline ≥30% during Part 1 and continued in Part 2. This outcome measure was pre-specified to collect data only for Part 2.
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 6 | 9
μmol/L | -488.19 (50.532) | 4.03 (46.496)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -492.23, 95% CI 2-sided [-614.59 to -369.87], Standard Error of Mean 55.588

12. Other Pre Specified Outcome: Part 2 Double-blind Phase: Percent Change From Baseline in Blood Phe Level to Weeks 5 and 6 (Averaged Over a 2-week Period) in Classical PKU Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: as for outcome 11
Time Frame: Baseline, Weeks 5 and 6 (average of the 2-week period)
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Part 2: Sepiapterin | Part 2: Placebo
Number analyzed (Participants) | 6 | 9
percent change | -55.83 (9.182) | 18.90 (8.286)
Statistical Analysis 1: Comparison: Part 2: Sepiapterin vs Part 2: Placebo; Test type: Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -74.73, 95% CI 2-sided [-97.72 to -51.74], Standard Error of Mean 10.436

13. Other Pre Specified Outcome: Part 1 Open-label Run-in Phase: Mean Change From Baseline (Part 1) in Blood Phe Level to Weeks 1 and 2 (Averaged Over a 2-week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: Baseline was defined as the average of Day -1 and Day 1 predose blood Phe levels in Part 1 Open-label Run-in Phase, and mean level at Weeks 1 and 2 was calculated as the average of blood Phe levels collected during the Week 1-2 analysis visit window. LS mean and SE were calculated using MMRM method.
Time Frame: Baseline (Part 1), Weeks 1 and 2 (average of the 2-week period)
Population: FAS included all participants who were enrolled and received at least 1 dose of open-label study drug in Part 1. Here "Overall number of participants analyzed" = participants of FAS with Phe reduction from Baseline ≥30% during Part 1.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Part 1: Sepiapterin
Number analyzed (Participants) | 103
μmol/L | -462.17 (203.620)

14. Other Pre Specified Outcome: Part 1 Open-label Run-in Phase: Percent Change From Baseline (Part 1) in Blood Phe Level to Weeks 1 and 2 (Averaged Over a 2-week Period) in Participants With Phe Reduction From Baseline ≥30% During Part 1
Description: as for outcome 13
Time Frame: Baseline (Part 1), Weeks 1 and 2 (average of the 2-week period)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: Sepiapterin
Number analyzed (Participants) | 103
percent change | -65.25 (15.764)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 42
Description: Safety analysis set included all participants who received at least 1 dose of study drug, including during Part 1.
Arm/Group | Part 1: Sepiapterin | Part 2: Sepiapterin | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/56 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 15/157 | 14/56 | 11/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Sepiapterin (N=157) | Part 2: Sepiapterin (N=56) | Part 2: Placebo (N=54)
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT05099640/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT05099640/SAP_001.pdf